CLINICAL TRIAL: NCT03291990
Title: A Pilot Study to Assess Feasibility of 5 Fraction Hypofractionated Stereotactic Radiosurgery Along With Standard Temozolomide as a Lymphocyte Sparing Therapy for Glioblastoma Multiforme
Brief Title: 5 Fraction Stereotactic Radiosurgery With Temozolomide for Glioblastoma Multiforme
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J1745; IRB00129314 (Other: JHMIRB)
Record Dates: First submitted 2017-09-15; First posted 2017-09-25 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-02

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: 5 fraction hypofractionated stereotacic radiosurgery along with standard temozolomide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5 fraction radiotherapy with standard temozolomide (Experimental): 5 fraction hypofractionated stereotactic radiosurgery along with standard temozolomide
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 5 fraction hypofractionated stereotactic radiosurgery along with standard temozolomide
  Other Names: 5 fraction radiosurgery with temozolomide

SUMMARY:
This investigation is not only to develop an improved radiation/temozolomide approach, but also develop a regimen with potential to form the basis of better combined therapy with immune based treatments.

DETAILED DESCRIPTION:
Glioblastoma has a poor prognosis with median survival is 14-16 months for patients enrolling in clinical trials, and across the United States one year survival is reported in the Surveillance, Epidemiology, and End Results (SEER) registry to be only 35%. Radiation treatment related lymphopenia has been associated with poor tumor outcome in Glioblastoma and a variety of other tumor types. As this lymphopenias is prolonged, it may also reduce efficacy of the checkpoint inhibitor lymphocyte mediated immune therapies now approved by the FDA for an increasing number of indications. Modeling and clinical studies suggest that administering radiation over 5 or fewer days (rather than standard 30 days of treatment) may reduce the incidence of lymphopenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age.
* Patients must have confirmed glioblastoma multiforme (GBM)
* Maximum postoperative dimension of cavity plus residual contrast enhancing tumor of < * If a patient is found on the radiation planning scan to have a tumor target larger than this size, the patient will be removed from the study.
* Patient must be selected for standard temozolomide chemotherapy to be administered with radiotherapy.
* Patient agrees to have 10 week follow-up visit at a participating Johns Hopkins facility.
* Patient agrees to allow access to or provide clinical, imaging, and laboratory follow-up information for three years whether or not obtained from Johns Hopkins providers.

3.1.7. Patients must not have received prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agents (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, Tumor-infiltrating lymphocytes (TIL), Lymphokine-Activated Killer Cell (LAK) or gene therapy), or hormonal therapy for their brain tumor. Glucocorticoid therapy is allowed.

* Patients must have a Karnofsky performance status 60% or higher (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Patients must be able to provide written informed consent.
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test.
* Patients must be able to undergo MRI scan with gadolinium contrast for treatment planning.

Exclusion Criteria:

* Patients may not plan to receive any other approved or investigational agents to treat their glioblastoma besides temozolomide prior to the evaluation visit 10 weeks after the initiation of radiotherapy and temozolomide.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, or other cancer from which the patient has been disease free for at least 2 years.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements will be excluded.
* Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and up to 12 weeks after the study are excluded. This applies to any woman who has not experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months). Male subjects must also agree to use effective contraception for the same period as above.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Rate of change of lymphopenia | 10 weeks
  To measure the incidence of > grade 3ymphopenia resulting from combined stereotactic hypofractionated radiotherapy and standard temozolomide in malignant glioma at the the standard follow-up 10 weeks after the initiation of therapy.

SECONDARY OUTCOMES:
Percentage change in Cluster of differentiation 4 (CD4) count (antigen found on helper T cells) | 10 weeks
  To describe the percent of patients with CD4 count < 200 mm/m3 at the standard week 10 follow-up
Rate of change of lymphocytes | 10 weeks
  Describe recovery of lymphocyte counts during routine clinical follow-up.
Rate of survival | 10 weeks
  To describe clinical/survival outcome based upon routine standard of care.
Rate of change in serious adverse events | 10 weeks
  To describe treatment related serious adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kleinberg, MD, Principal Investigator — SKCCC at Johns Hopkins (East Baltimore)
Locations (3):
- United States (3):
  - Sibley Hospital, Washington D.C., District of Columbia
  - Suburban Hospital, Washington D.C., District of Columbia
  - SKCCC at Johns Hopkins (East Baltimore), Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No